CLINICAL TRIAL: NCT05538702
Title: Acute Oral Effects of Heated Tobacco Products Compared to Traditional Cigarettes
Brief Title: Acute Oral Effects of Heated Tobacco Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 91-3/2015
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Nicotine Dependence, Cigarettes
Keywords: nicotine; heated tobacco product; blood flow; cigarette
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Heated tobacco product with bland taste unit (Experimental): Nicotine content: 0,5 mg
  Interventions: Device: IQOS 3.0 DOU with bland taste unit (Heated Tobacco Product)
- Heated tobacco product with menthol taste unit (Experimental): Nicotine content: 0,5 mg
  Interventions: Device: IQOS 3.0 DUO with menthol taste unit (Heated Tobacco Product)
- Conventional cigarette (Experimental): Nicotine content: 0,5 mg
  Interventions: Device: Marlboro Gold (Conventional cigarette)
- Heated tobacco product turned off with a bland taste unit (Placebo Comparator): Placebo device
  Interventions: Device: IQOS 3.0 DUO turned off with a bland taste unit

INTERVENTIONS:
Device: IQOS 3.0 DOU with bland taste unit (Heated Tobacco Product) — Heated tobacco products (HTP) are devices which heat but do not burn tobacco. They do not produce cigarette smoke but rather an aerosol.
  Other Names: IQOS 3.0 DUO; HEETS Bronze Selection
  Arms: Heated tobacco product with bland taste unit
Device: IQOS 3.0 DUO with menthol taste unit (Heated Tobacco Product) — Heated tobacco products (HTP) are devices which heat but do not burn tobacco. They do not produce cigarette smoke but rather an aerosol.
  Other Names: IQOS 3.0 DUO; HEETS Blue Selection
  Arms: Heated tobacco product with menthol taste unit
Device: Marlboro Gold (Conventional cigarette) — Conventional cigarette
  Other Names: Marlboro Gold 0,5 mg
  Arms: Conventional cigarette
Device: IQOS 3.0 DUO turned off with a bland taste unit — Placebo device
  Other Names: IQOS 3.0 DUO; HEETS Bronze Selection
  Arms: Heated tobacco product turned off with a bland taste unit

SUMMARY:
Heated tobacco products (HTP) are devices which heat, but not burn tobacco. They do not produce cigarette smoke but rather an aerosol. HTPs are marketed as less harmful alternatives to smoking. Use and awareness of these devices have grown exponentially in recent years, with probably millions of people currently using them. There is very little literature about them, so it is quite important to study the effects caused on the human body by these products.

The benefits and risks of HTP use are uncertain. There is no research on the acute oral effects of HTPs in the scientific literature.

DETAILED DESCRIPTION:
Measurements of acute oral effects before and after using HTP with bland flavour (HEETS Bronze Selection), with methol flavour (HEETS Blue Selection), conventional cigarette and placebo device:

measurement of exhaled CO changes by Smokerlyzer piCO measurement of oral mucosal blood flow changes by Perilam PSI System High Resolution (LASCA method) measurement of blood pressure and pulse by an automatic blood pressure monitor (Omron M2, Omron Healthcare Inc., Kyoto, Japan)

ELIGIBILITY:
Inclusion Criteria:

* age: 18-49 years
* signed consent form
* smoking regularly heated tobacco product and/or conventional cigarette for > half year

Exclusion Criteria:

* not pregnant and not planning pregnancy in the next 6 month BMI index < 30
* no severe parodontal disease
* no acute illness in the last 2 weeks
* no chronic disease (eg.: diabetes)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline in blood flow after smoking | baseline, immediately after smoking, and 15 minutes after smoking
  The blood flow changes are measured by Laser Speckle Contrast Analyzer (LASCA) before (baseline), immediately after, and 15 minutes after smoking.

CONTACTS AND LOCATIONS:
Locations (1):
- Semmelweis University, Department of Prosthodontics, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Undecided